CLINICAL TRIAL: NCT04245254
Title: GutMe!: IBS and Collagen Protein Powder an Interventional Study
Acronym: GutMe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProofPilot (Industry)
Collaborators: Qina (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2329
Record Dates: First submitted 2020-01-25; First posted 2020-01-28 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Irritable Bowel Syndrome; Irritable Bowel; Irrit
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Single arm interventional study.
Masking Description: All participants receive one brand of collegen protien powder
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Single arm study. Receives collagen protein powder.
  Interventions: Dietary Supplement: Collagen Protien Powder

INTERVENTIONS:
Dietary Supplement: Collagen Protien Powder — Collegen Protein Powser

SUMMARY:
In this study we would like to understand how or if a food-based supplement affects gut symptoms such as bloating, stomach cramps and irregular bowel habits. Through using a digital symptom tracking app for a few weeks, you may just learn more about exactly what is triggering your symptoms!

ELIGIBILITY:
Inclusion Criteria:

* US based
* self report bloating

Exclusion Criteria:

* vegan or vegetarian diet
* suffering from any skin disorders
* kidney disease
* treated medical issues
* glutamine sensitivity

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women are more affected by IBS than men.
Enrollment: 50 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in self-reported IBS symptoms | Baseline, Week 4 and Week 10

CONTACTS AND LOCATIONS:
Locations (1):
- ProofPilot (Virtual Study: https://p.proofpilot.com), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to make PID available to other researchers.

REFERENCES:
- [Derived] Abrahams M, O'Grady R, Prawitt J. Effect of a Daily Collagen Peptide Supplement on Digestive Symptoms in Healthy Women: 2-Phase Mixed Methods Study. JMIR Form Res. 2022 May 31;6(5):e36339. doi: 10.2196/36339. PMID 35639457